CLINICAL TRIAL: NCT00216164
Title: Phase II Study of Rituximab and Gemcitabine in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma: Hoosier Oncology Group LYM03-64
Brief Title: Rituximab and Gemcitabine for Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of response at the first efficacy analysis
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Eli Lilly and Company (Industry); Walther Cancer Institute (Other)
Responsible Party: Michael Robertson, M.D., Hoosier Oncology Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG LYM03-64
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Lymphoma, B-Cell
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma | interventions — Rituximab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Rituximab + Gemcitabine for Relapsed or Refractory Diffuse Large B-Cell Lymphoma
  Interventions: Drug: Rituximab; Drug: Gemcitabine

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2, day 1 of 21 day cycle
Drug: Gemcitabine — Gemcitabine 1000 mg/m2, days 1 and 8 of 21 day cycle

SUMMARY:
Rituximab has been demonstrated to sensitize drug-resistant NHL cells to the cytotoxic actions of several chemotherapy agents by enhancing sensitivity of tumor cells to chemotherapy-induced apoptosis. Gemcitabine, a nucleoside analog that is used in several other malignancies, has shown very promising activity in patients with refractory Hodgkin's disease and low-grade NHL. The combination of rituximab and gemcitabine may have synergistic cytotoxic action in patients with relapsed or refractory DLBCL and possibly lead to improved response rates and demonstrable clinical benefit.

This trial will investigate the efficacy the combination of rituximab and gemcitabine in treating patients with relapsed or refractory DLBCL.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Rituximab 375 mg/m2 day 1 of 21 day cycle
* Gemcitabine 1000 mg/m2 days 1 and 8 of 21 day cycle

Subgroup 1. Relapsed after responding to first line chemotherapy, who are not candidates for salvage high-dose chemotherapy.

Subgroup 2. Failure to achieve a complete response or relapsed after responding to salvage chemotherapy (any number of salvage regimens allowed), who are not candidates for high-dose chemotherapy.

Subgroup 3. Refractory to first line chemotherapy and/or 1 (one) salvage chemotherapy regimen.

Subgroup 4. Progression after high-dose chemotherapy. Patients with progressive disease within 3 months of high-dose chemotherapy are not allowed.

Performance Status: ECOG performance status 0, 1, 2

Life expectancy: Not specified

Hematopoietic:·

* ANC ≥ 1,000/mm3·
* Platelets ≥ 100,000/mm3

Hepatic:·

* Total bilirubin ≤ 2.0 x ULN·
* ALT and AST ≤ 3 x ULN unless lymphoma involves the liver on CT scan then AST and ALT can be < 5 x ULN

Renal:·

* Serum creatinine ≤ 2.0 mg/dl (except for patients on dialysis)

Cardiovascular:·

* Not specified

Pulmonary:·

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven DLBCL which meet the criteria of any of the 4 subgroups
* Transformed DLBCL from a previous indolent NHL which meet the criteria of any of the 4 subgroups and have received at least one standard chemotherapy regimen for aggressive NHL or a biopsy upon progression of disease has been obtained to confirm the presence of DLBCL. The concomitant presence of a component of low grade lymphoma will NOT exclude participation
* Measurable disease per Standardized Response Criteria for Non-Hodgkin's Lymphoma
* Prior gemcitabine therapy is allowed.
* Negative pregnancy test

Exclusion Criteria:

* No history of life-threatening reactions to rituximab.
* No history of gemcitabine intolerance; prior gemcitabine therapy is allowed.
* No history of malignancy in the last 5 years (basal cell carcinoma of the skin excluded).
* No central nervous system or cerebrospinal fluid involvement
* No other investigational drugs received within 30 days prior to being registered for protocol therapy.
* No active infections.
* No current breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
· Evaluate response rates to the rituximab plus gemcitabine treatment combination in patients with relapsed or refractory DLBCL. | 18 months

SECONDARY OUTCOMES:
· Evaluate toxicity, time to progression and overall survival. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Robertson, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (9):
- United States (9):
  - Elkhart Clinic, Elkhart, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Center for Cancer Care, Inc., P.C., New Albany, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - AP&S Clinic, Terre Haute, Indiana

REFERENCES:
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/